CLINICAL TRIAL: NCT03211273
Title: A Prospective, Observational Study to Investigate Longterm Courses, Patterns, Determinants and State of Treatment of Cancer-related Fatigue in Germany (LIFT)
Brief Title: Longitudinal Investigation of Cancer-related Fatigue
Acronym: LIFT
Status: Withdrawn | Type: Observational
Why Stopped: no funding
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Other Study IDs: LIFT
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cancer-related Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Diurnal saliva samples (5 samples distributed over a day)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: Newly diagnosed breast, ovarian or colon cancer patients recruited 6 months post-diagnosis and followed up to 5 years post-diagnosis. No intervention.

SUMMARY:
In the LIFT study 2000 cancer patients will be recruited at 6 months after diagnosis and extensively surveyed over five years on factors that are associated with fatigue.

DETAILED DESCRIPTION:
The LIFT study aims to comprehensively investigate characteristics, determinants, and long-term course of fatigue. In addition, information shall be gained on the current state of fatigue treatment and care in Germany and on the needs of affected patients.

Data will be collected by mailed or online questionnaires at 6, 9, and 12 months as well as 2, 3, 4 and 5 years post-diagnosis from 2000 cancer patients. Besides questionnaires on socio-demographic, clinical and patient reported outcomes, saliva samples will be collected in order to gain new insights into biological mechanisms. Moreover, detailed data on screening, diagnosis and counseling as well as therapies offered and administered to reduce fatigue will be surveyed, as well as the patients' state of knowledge, perception and prevailing needs regarding fatigue. Tumor and cancer therapy data will be extracted from the Epidemiological Cancer Registry.

The results of the LIFT study aim to contribute to an improved, evidence-based and individualized treatment to avoid and ease cancer-related fatigue and will further promote patient-oriented offers and treatments.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosed with a primary tumor of breast, ovarian, or colon cancer
* Time since first diagnosis is 4 - 6 months
* Having received or currently receiving at least one of the following treatments: surgery, chemotherapy, radiotherapy, hormone therapy, or immune therapy.
* Able to understand and follow the study protocol.

Exclusion Criteria:

• Any additional malignant or unclear neoplasm or carcinoma in situ at or since time of diagnosis of the considered primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with breast, ovarian or colon cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity | from diagnosis to 1 year post-diagnosis
  assessed by EORTC QLQ-FA12 (European Organisation for Research and Treatment of Cancer Quality of Life Fatigue Questionnaire)
Impact of fatigue | from diagnosis to 1 year post-diagnosis
  assessed by the Brief Fatigue Inventory (BFI)
State of fatigue management | from diagnosis to 1 year post-diagnosis
  Questionnaire assessing the adherence to the National Comprehensive Cancer Network (NCCN) guidelines regarding management of cancer-related fatigue

SECONDARY OUTCOMES:
Quality of life functions and symptoms | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed by EORTC QLQ-C30
Sleep problems | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed by Pittsburgh Sleep Quality Index (PSQI)
Depression | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed by Patient Health Questionnaire (PHQ-9)
Body mass index | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  calculated from weight and height
Total physical activity | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed by a questionnaire regarding walking, cycling, and exercise behavior
Diurnal cortisol rhythm | 1 year post-diagnosis
  assessed in saliva
Return to work | 6, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed by a questions regarding occupational issues
Hot flashes | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed only for women
Anxiety | 6, 9, 12 months and 2, 3, 4, and 5 years post-diagnosis
  assessed by the Generalized Anxiety Disorder Questionnaire (GAD-7)

IPD SHARING:
Plan to Share IPD: Undecided